CLINICAL TRIAL: NCT04339166
Title: A Multicenter Clinical Study on Embryo Selection by Using the Ploidy of Cell Free DNA in Embryo Culture Medium
Brief Title: Embryo Selection by Noninvasive Preimplantation Genetic Test
Acronym: ESNi-PGT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University Third Hospital (Other)
Collaborators: Jinling Hospital, China (Other); Reproductive Medical Center of Hebei Maternity Hospital (Unknown); Northwest Women's and Children's Hospital, Xi'an, Shaanxi (Other); The First Medical Center of Chinese People's Liberation Army General Hospital (Unknown); Shengjing Hospital (Other); First Affiliated Hospital, Sun Yat-Sen University (Other); Reproductive & Genetic Hospital of CITIC-Xiangya (Other); Yikon Genomics Company, Ltd (Unknown); Peking University Shenzhen Hospital (Other); The Second Hospital of Hebei Medical University (Other); West China Second University Hospital (Other); Second Affiliated Hospital of Wenzhou Medical University (Other); Third Affiliated Hospital of Zhengzhou University (Other)
Responsible Party: Principal Investigator, Jie Qiao, Professor, Peking University Third Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: ESNi-PGT
Record Dates: First submitted 2020-04-01; First posted 2020-04-09 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Infertility; Chromosome Abnormality
Keywords: Culture media; Embryonic cell-free DNA; Euploidy
MeSH Terms: conditions — Infertility; Chromosome Aberrations

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Single thawed blastocyst transfer with blastocyst selection according to the analysis of NICS and morphologic score.
  Interventions: Diagnostic Test: Non-invasive chromosome screening（NICS）
- Group B (No Intervention): Single thawed blastocyst transfer with blastocyst selection according to morphologic score.

INTERVENTIONS:
Diagnostic Test: Non-invasive chromosome screening（NICS） — NICS is noninvasive chromosome screening approach to analysis the euploidy by free DNA in embryo culture medium
  Arms: Group A

SUMMARY:
The objective of this study is to explore whether non-invasive chromosome screening (NICS) can be used as an effective indicator for embryos selection besides morphology through a multicenter randomized controlled trial, by comparing the differences of live birth rate, pregnancy rate and miscarriage rate between the two groups of embryo selection by "NICS+ morphology" and embryo selection only by "morphology" in IVF cycle.

DETAILED DESCRIPTION:
Chromosomal abnormalities commonly exist in early human embryos, and often cause embryo implantation failure and pregnancy loss in in-vitro fertilization (IVF) treatments. Preimplantation genetic testing for aneuploidies (PGT-A) by comprehensive chromosome screening (CCS) has been widely applied in IVF practices to select embryos with normal ploidy. Although multiple clinical trials have demonstrated improved clinical outcomes with PGT-A, it's in controversial for whether PGT-A is truly worthwhile to be offered to all IVF patients. One of the main concerns is that it involves an embryo biopsy procedure, which is invasive and the long-term safety issue of the embryo biopsy remains to be fully investigated.

In recent years, researchers have found that the spent medium of embryo culture contains trace amount of cell-free DNA, which may reflect the ploidy of the embryo. The non-invasive chromosome screening (NICS) approach utilizing spent culture medium samples has been evaluated in studies. However, the clinical value of NICS as a new effective indicator to evaluate embryo competence so far has not been justified by randomized clinical trials.

The main purpose of this project is to verify whether NICS can be used as a new effective indicator for evaluating embryo developmental potential through multi-center, randomized clinical trials

ELIGIBILITY:
Inclusion Criteria:

1. Infertile couples receiving IVF- ICSI procedure for assisted reproduction cycle
2. Female age: 35 - 42 years old
3. Women receiving controlled ovarian hyperstimulation treatment (including ultra-long protocol、long-protocol 、short protocol treatment with GnRH agonist and GnRH antagonist treatment protocol); and the number of oocytes ≥6; The female BMI is from 18 to 30kg/m2.
4. Culture embryos to blastocyst stage and all the blastocysts will be single cryopreserved.
5. Single frozen-thawed blastocyst Transferred for the first time
6. The number of blastocysts ≥2, morphology grade (above 4BC/4CB)
7. Written informed consent

Exclusion Criteria:

1. One of couples with IVF or ICSI contraindications(such as poorly controlled type I or type II diabetes; liver disease or dysfunction; kidney disease or renal function abnormality; significant anemia; history of deep venous thrombosis, pulmonary embolus; history of cerebrovascular accident; uncontrolled hypertension or diagnosed heart disease; history of cervical, endometrial or breast cancer; undiagnosed vaginal bleeding.)
2. PGT cycles
3. Women who have pathologies or malformations that affect the pregnancy outcome: genital malformations, untreated hydrosalpinx, untreated uterine infections, intramural myomas > 4cm , benign tumor of pelvic and abdominal cavity> 4cm, intimal thickness<8mm, pituitary tumors and malignant tumors of various tissues and organs during the patient's participation in the study
4. Untreated hyperprolactinemia, thyroid disease, adrenal disease
5. Women with endometrial polyps that were not treated before embryo transfer

Ages: 35 Years to 42 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — IVF patients
Enrollment: 1152 (Actual)
Dates: Start 2020-04-16 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-08-06 (Actual)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after the first embryo transfer
  Number of women with ongoing pregnancies after the first transfer/ number of women randomized to the specific group

SECONDARY OUTCOMES:
Clinical pregnancy rate | 7 weeks after the first embryo transfer
  Number of women with clinical pregnancies after the first transfer / number of women randomized to the specific group
Miscarriage rate | Miscarriage：28 weeks of after the first embryo transfer； First trimester miscarriage(early miscarriage)：12 weeks of after the first embryo transfer；
  Number of pregnancy losses / number of clinical pregnancies after the first transfer.
Live birth rate | within 2 weeks after live birth
  Number of women with live births after the first transfer / number of women randomized to the specific group.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Qiao, Principal Investigator — Peking University Third Hospital
Locations (13):
- China (13):
  - The First Affiliated Hospital,Sun Yat-sen University, Guanzhou, Guangdong
  - Peking University Shenzhen Hospital, Shenzhen, Guangdong
  - Hebei Maternity and Reproductive hospital, Shijiazhuang, Hebei
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The Third Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Reproductive & Genetic Hospital of Citic-Xiangya, Changsha, Hunan
  - Jinling Hospital,Nanjing University,School Medicine, Nanjing, Jiangsu
  - Shengjing Hospital of China Medical University, Shenyang, Liaoning
  - West China Second Hospital of Sichuan University, Chengdu, Sichuan
  - The Second Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
  - Peking University Third Hospital, Beijing
  - The First Medical Center of Chinese People's Liberation Army General Hospital, Beijing
  - Northwest women's and children's hospital, Xi'an

IPD SHARING:
Plan to Share IPD: Yes
Data may be shared with proper internal and ethical approval. De-identified data may also be shared with approved study investigators.
Supporting Information: Study Protocol
Time Frame: After the study has been completed
Access Criteria: Proper internal and ethical approval; protect patient confidentiality; approve by study investigators

REFERENCES:
- [Derived] Huang J, Rong L, Zeng L, Hu L, Shi J, Cai L, Yao B, Wang XX, Xu Y, Yao Y, Wang Y, Zhao J, Guan Y, Qian W, Hao G, Lu S, Liu P, Qiao J. Embryo selection through non-invasive preimplantation genetic testing with cell-free DNA in spent culture media: a protocol for a multicentre, double-blind, randomised controlled trial. BMJ Open. 2022 Jul 27;12(7):e057254. doi: 10.1136/bmjopen-2021-057254. PMID 35896299